CLINICAL TRIAL: NCT05062317
Title: Risk-Stratified Adjuvant Therapy: ctDNA-Directed Post-Hepatectomy Chemotherapy for Patients With Resectable Colorectal Liver Metastases
Brief Title: ctDNA-Directed Post-Hepatectomy Chemotherapy for Patients With Resectable Colorectal Liver Metastases
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021-0584
Record Dates: First submitted 2021-09-21; First posted 2021-09-30 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Liver Metastases
MeSH Terms: interventions — Leucovorin; Fluorouracil; Oxaliplatin; Irinotecan; Capecitabine; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ctDNA (Low Risk) (Experimental): Will receive less intense chemotherapy, such as capecitabine or 5-fluorouracil.
  Interventions: Drug: Leucovorin; Drug: Capecitabine
- ctDNA (High Risk) (Experimental): Will receive more intense chemotherapy. This may include resuming the chemotherapy you received before surgery (for example, FOLFOX [5-fluorouracil, leucovorin and oxaliplatin] or FOLFIRI [5-fluorouracil, leucovorin and irinotecan] with or without bevacizumab)
  Interventions: Drug: Leucovorin; Drug: 5-FLUOROURACIL; Drug: Oxaliplatin; Drug: Irinotecan; Drug: Capecitabine; Drug: Bevacizumab

INTERVENTIONS:
Drug: Leucovorin — Given by PO
  Other Names: Citrovorum; Wellcovorin®
Drug: 5-FLUOROURACIL — Given by IV
  Arms: ctDNA (High Risk)
Drug: Oxaliplatin — Given by PO
  Other Names: Eloxatin
  Arms: ctDNA (High Risk)
Drug: Irinotecan — Given by IV
  Arms: ctDNA (High Risk)
Drug: Capecitabine — Given by IV
  Other Names: Xeloda
Drug: Bevacizumab — Given by IV
  Other Names: Avastin™; Anti-VEGF monoclonal antibody; rhuMAb-VEGF
  Arms: ctDNA (High Risk)

SUMMARY:
To determine if the detection of ctDNA after surgical resection of CLM can stratify patients into high and low-risk cohorts for early disease recurrence in order to inform post-operative adjuvant therapy.

DETAILED DESCRIPTION:
Primary Objective:

• To assess 1-year recurrence-free survival rate following liver resection of CLM with curative intent among ctDNA-negative patients who receive risk-stratified postoperative chemotherapy

Secondary Objectives:

* To assess recurrence-free survival following liver resection of CLM with curative intent among ctDNA-positive patients
* To assess overall survival following liver resection among ctDNA-negative and ctDNA-positive patients
* To evaluate the proportion of ctDNA-negative at 1-year post-resection
* To compare survival of ctDNA-negative patients undergoing ctDNA-guided postoperative chemotherapy to historical controls
* To evaluate proportion of patients in each arm who change chemotherapy in response to ctDNA measurement
* To delineate the pattern of disease recurrence
* To assess ctDNA sensitivity and specificity for predicting disease recurrence
* To evaluate MDASI-GI during the course of postoperative therapy
* To evaluate and correlate patient molecular subtypes and characterization of tumor biologic factors that are associated with ctDNA detection
* To evaluate surgery-related adverse events occurring up to 90 days after surgery, and chemo-related adverse events occurring up to 30 days after the last dose of chemotherapy

Outcome Measures:

Primary:

• Recurrence-free survival at 1-year post-hepatectomy among ctDNA-negative patients

Secondary:

* Recurrence-free survival at 1-year post-hepatectomy among ctDNA-positive patients
* Overall survival (OS) among ctDNA-negative and ctDNA-positive patients
* ctDNA-negativity at 1-year post-resection
* Proportion of patients in each group with chemotherapy regimen change in response to ctDNA dynamics
* Pattern of disease recurrence (i.e., liver, systemic, salvageable vs. unsalvageable)
* ctDNA sensitivity/specificity for recurrent disease overall by timepoint
* MDASI-GI at clinic visits during course of postoperative therapy
* Tumor radiologic, histologic, and molecular profiling and correlative characterization based upon ctDNA detection
* Adverse events

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥18 years of age with CLM undergoing elective hepatectomy with curative intent (primary colorectal primary cancer previously removed OR being removed at time of hepatectomy) after preoperative chemotherapy (i.e., FOLFOX/FOLFIRI +/- bevacizumab or panitumumab/cetuximab) from 07/01/2021 - 12/31/2023
* Must receive ≥ 4 cycles of preoperative chemotherapy

Exclusion Criteria:

* Patients with primary colorectal tumor that will remain in situ
* Inability to undergo postoperative chemotherapy, or postoperative chemotherapy not planned a priori
* Unwilling/unable to undergo blood draws for ctDNA, patient or provider-determined
* Other active malignancies requiring treatment
* Women who are pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-04-26 (Actual); Primary Completion 2027-02-28 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
To establish the 1-year recurrence-free survival rate following liver resection of CLM with curative intent among ctDNA-negative patients who receive risk-stratified postoperative chemotherapy | through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Newhook, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center website — http://www.mdanderson.org